CLINICAL TRIAL: NCT00951509
Title: Computer-based and Virtual Assessment of Power Wheelchair Mobility
Brief Title: Virtual Reality Based Testing of Power Wheelchair Driving Skills
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: A6035-R; 02691 (Other: VAPHS IRB)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Results first posted 2015-08-24 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-07

CONDITIONS: Spinal Cord Injury; Spina Bifida; Spinal Cord Disease
Keywords: Electric power wheelchair driving; rehabilitation; driving assessments
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Dysraphism; Spinal Cord Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Condition 1 (PC Screens with No Rollers): All subjects (Repeated - measures study design): All subjects were evaluated with the Power Mobility Road Test (PMRT).
  Interventions: Other: Power Mobility Road Test (PMRT)
- Condition 2 (PC Screens with Rollers): All subjects (Repeated - measures study design): All subjects were evaluated with the Power Mobility Road Test (PMRT).
  Interventions: Other: Power Mobility Road Test (PMRT)
- Condition 3 (VR Screens with No Rollers): All subjects (Repeated - measures study design): All subjects were evaluated with the Power Mobility Road Test (PMRT).
  Interventions: Other: Power Mobility Road Test (PMRT)
- Condition 4 (VR Screens with Rollers): All subjects (Repeated - measures study design): All subjects were evaluated with the Power Mobility Road Test (PMRT).
  Interventions: Other: Power Mobility Road Test (PMRT)
- Condntion 5 (Real-world driving): All subjects (Repeated - measures study design): All subjects were evaluated with the Power Mobility Road Test (PMRT).
  Interventions: Other: Power Mobility Road Test (PMRT)

INTERVENTIONS:
Other: Power Mobility Road Test (PMRT) — All subjects will underwent the Power Mobility Road Test (PMRT), and the clinicians scored the driving performance within each condition.

SUMMARY:
The purpose of this research study is to examine whether computer based or virtual reality based driving assessments are as useful as real-world power wheelchair driving tests in measuring driving performance and whether they may be useful in helping to identify the problems that some individuals may have with driving power wheelchairs. The specific aims are as follows:

Specific Aim 1: To develop computer-based and VR-based wheelchair driving assessments for both drivers and non-drivers that correspond to an accepted real-world driving assessment (Power Mobility Road Test) and compare them to the real-world assessment and to each other.

Specific Aim 2: To develop additional features of the computer-based and VR-based assessments that present dynamic tasks and determine whether skills on these tasks can be delineated within the virtual environment.

DETAILED DESCRIPTION:
This study has an experimental, repeated measures design with validity and reliability testing. In Phase 1 of the study, we designed and developed the software needed to deliver the computer-based and VR-based testing environments. In Phase 2 of the study, we improved on the design iterations of Phase I, recruited a sample of 31 Electric Power wheelchair (EPW) users and delivered the simulator based driving assessment using a pool of clinicians to assess the reliability of system in real world and in the virtual environments.

Phase II: Research Protocol:

Experimental Set-up:

VRSIM consisted of two display options, three 6' X 8' back projected screens (field of view 160°) (VR screens) and a single 22" desktop monitor (field of view 90°) (PC screens), both with the first-person perspective viewpoint (Fig.1). The virtual environment consisted of a simulation of an indoor office space with a kitchen; a lounge area and set of hallways lined by offices, and incorporated the tasks of the PMRT (Fig.2). Participants interacted with VRSIM either using dual rollers that interfaced with drive wheels of the wheelchair ('Rollers ON' driving mode) or using an instrumented wheelchair joystick through a custom software ('Rollers OFF' driving mode). The custom software uses a proportional derivative mathematical model to simulate the real-world motion of the EPW within the virtual environment. VRSIM was designed with two display options and two user input modalities to assess the feasibility of using such a system with different interfaces in different settings, such as in a busy wheelchair clinic (using the much immersive VR screens with rollers) or in a user's home (with the user's personal computer and the customized joystick).

The "actor/driver" in the VRSIM was a virtual model of a person sitting in a standard commercially available EPW power wheelchair (width 0.671 m, length 0.701 m). A horizontal slider bar that indicated the real time location of the virtual wheelchair with respect to virtual obstacles was added to this version (Fig.1, 2). This helped display warnings when the chair was too close to obstacles, especially when the obstacles were behind the driver. Participants were expected to drive along the course indicated by arrows touching or passing through preset milestone markers signified by semi-transparent balloons. These sequentially displayed milestones defined the tasks of the virtual PMRT. Participants were instructed to complete every task as quickly and accurately as possible. An equivalent PMRT driving course was charted out in an office space for the real world driving evaluation.

Data collection:

After informed consent, participants performed up to 2 practice sessions within the virtual driving course. Participants reported their level of comfort and sense of being in control in the VRSIM during practice based on which a value between 1.0 and 4.0 was selected for the linear and angular speed gains in VRSIM. In addition, participants were asked to select a different pre-programmed driving profile on their wheelchairs (e.g. "indoor" profile), which was similar to their everyday driving profile to obtain optimum driving speed. Optional breaks for 5-10 minutes were provided between driving sessions. For both the PC and VR screens, participants drove through the complete driving course: two trials with the Rollers ON driving mode, one trial with the Rollers OFF driving mode, and one trial in the real-world PMRT driving course constituted to a total of 5 driving conditions (Table 1). A balanced randomization scheme was used to set the order of the five driving conditions.

From a group of 6 clinicians comprised of 1 occupational therapist, 3 physical therapists, and 2 physicians, 2 clinicians were randomly assigned as the evaluation team for each participant. The team always had 1 certified Assistive Technology Professional with more than 5 years of experience in power wheelchair driving evaluations. The assigned clinicians independently scored every PMRT task during all the driving trials using the following criteria: 4: completed independently, 3: completed hesitantly requiring several trials and minor accidents, 2: commits serious accidents that may cause harm to driver or other people, 1: unable to complete a task. Each clinician had a separate PMRT scoring sheet for each trial.

Repeat Testing:

Subjects underwent all five testing scenarios twice, returning on a second visit in no earlier than 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between 18 to 80 years old.
* Subjects must have a diagnosis of SCI, spina bifida, syringomyelia, spinal stenosis, transverse myelitis, ALS, spinal cord disease, multiple sclerosis, stroke, polytraumatic injury, or TBI with residual motor, sensory, or cognitive impairments that impair mobility.
* Subjects must use a power wheelchair or an attendant propelled manual wheelchair for all or part of their mobility.
* Subjects must be able to provide informed consent.
* Subjects must have very basic cognitive, visual, and motor skills to interact with an interface.

Exclusion Criteria:

* Subjects who have active pelvic or thigh wounds. (They may be worsened by prolonged sitting).
* Subjects with a history of seizures in the last 90 days. (A computer screen task has the potential to induce seizures).
* Subjects who do not pass the screening protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with physical disabilities who have a mobility impairment due to any any spinal cord disease condition (e.g. Spinal Cord Injury, Spina Bifida)
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rory A. Cooper, PhD, Principal Investigator — Director, Center of Excellence for Wheelchairs and Related Technology
Locations (1):
- VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Institutional Review Boards of the Veteran Affairs Pittsburgh Healthcare System and the University of Pittsburgh approved the protocol for this research study. Participants were recruited at the 31st National Veterans Wheelchair Games (NVWG), VA Wheelchair clinic, and the UPMC Center of Assistive Technology.
Groups:
- Participants Who Qualified for the Study: All participants who qualified for the study, performed electric power wheelchair (EPW) driving under five driving conditions, while clinicians observed and assessed the EPW users' driving performance. The first four conditions were conducted in virtual environments (with different interfaces in each condition, as listed below) and condition 5 was conducted in the real world - Condition 1 - Desktop screens with no roller systems Condition 2- Desktop screens with roller systems Condition 3 - Immersive virtual reality screens with no roller systems Condition 4 - Immersive virtual reality screens with roller systems Condition 5 - Real world EPW driving
Period: Overall Study
Arm/Group | Participants Who Qualified for the Study
Started | 31
Driving Condition 1 | 29
Driving Condition 2 | 29
Driving Condition 3 | 25
Driving Condition 4 | 28
Driving Condition 5 | 30
Completed | 29
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Power Mobility Road Test (PMRT): All subjects were asked to complete the "real world" power mobility evaluation via the PMRT.
  Computer-Based Test: All subjects were asked to complete the computer-based evaluation designed to simulate real world driving in a 2D environment.
  Virtual Reality Test: All subjects were asked to complete the virtual-based evaluation designed to simulate real world driving in a 3D environment.
Arm/Group | All Subjects
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 15
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Composite Power Mobility Road Test (PMRT) Scores
Description: The computer-based and the virtual environments will be modeled after and scored similarly to the real world PMRT. The PMRT contains two domains: Structured Elements/Tasks and Unstructured Skilled Driving. The first domains contain 16 tasks that include activities such as passing through standard width doorways, and turning a ninety-degree turn, turning 180 degrees. In both domains, each task is scored from 1 to 4, depending on speed and the number of collisions that occur with obstacles. A total score for the entire test is calculated out of a possible 64 points, and the final score on the test reflects the percentage of total points acquired1. A passing score is a percentage of > 95%.
Time Frame: Baseline in-lab testing
Population: Majority of the participants (41%) had a spectrum of multiple disabilities ranging from stroke, spinal stenosis, osteoarthritis, emphysema, and cerebral degeneration, followed by 11 participants (35%) with spinal cord injury.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Condition 1; Condition 2; Condition 3; Condition 4; Condition 5: Power Mobility Road Test (PMRT): All subjects were evaluated using the PMRT in the five different conditions, and reliability was assessed using Intra-class Correlation (ICC) coefficients.There was no difference in the mean scores between the five different driving conditions.
Arm/Group | Condition 1 | Condition 2 | Condition 3 | Condition 4 | Condition 5
Number analyzed (Participants) | 29 | 29 | 25 | 28 | 30
units on a scale | 95.3 (5.4) | 96.09 (7.8) | 93.75 (7.03) | 96.88 (8.2) | 100 (1.56)

ADVERSE EVENTS:
Time Frame: Over the entire course of the study.
Groups:
- Power Mobility Road Test: With 12 structured tasks and 4 dynamic tasks, adding to a total of 16 tasks with a minimum score of 1 and maximum of 4 in each task, it is possible to score in the range of 16 - 64 during a driving trial. To assess the driving performance, the total score for each trial was calculated and expressed as a percentage, termed "Composite score". A Composite score of 95 % or greater would suggest that the user is a safe driver.
Arm/Group | Power Mobility Road Test
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No